CLINICAL TRIAL: NCT00750100
Title: Among ICSI Patients Undergoing Antagonist Protocols With Recombinant FSH, Does Replacement of Recombinant FSH by 200 IU of hCG in the Late Follicular Phase Compared With Continuing Recombinant FSH, Result in a Similar Number of Oocytes?
Brief Title: Low Dose hCG in the Late Follicular Phase
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Paul Devroey, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC REF 2006-157
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2008-09

CONDITIONS: Infertility
Keywords: infertility; IVF; hCG; primary infertility; secondary infertility; patients requiring in-vitro fertilisation
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; follitropin beta

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Patients undergo a standard antagonist protocol for in-vitro fertilisation, and are stimulated with recombinant gonadotropins.
  Interventions: Drug: recombinant gonadotropins
- B (Experimental): Patients are undergo an antagonist protocol for in-vitro fertilisation and are stimulated with recombinant gonadotropins. When the patient has an estradiol value of 600 ng/L or more and when the patient has at least 6 follicles of 12 mm, the administration of gonadotropins is stopped and replaced by low dose human chorionic gonadotropins.
  Interventions: Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin — hCG 200IU in the late follicular phase
  Other Names: Pregnyl, NV Organon, Oss, The Netherlands
  Arms: B
Drug: recombinant gonadotropins — 200 IU per day during controlled ovarian stimulation
  Other Names: Puregon, NV Organon, Oss, The Netherlands
  Arms: A

SUMMARY:
In this study,the investigators compared two protocols for controlled ovarian hyperstimulation in infertility patients requiring IVF. In the control group, the patient undergoes a standard antagonist protocol. In the study group, the administration of gonadotropins is stopped in the late follicular phase and replaced by low dose human chorionic gonadotropins. The primary endpoint of the study is the number of oocytes retrieved in both groups.

ELIGIBILITY:
Inclusion Criteria:

* < 36 years on day of randomisation
* FSH < 12 in the early follicular phase
* Normal ultrasound scan
* BMI between 18 and 29 (both inclusive)
* Randomisation at outpatient clinic

Exclusion Criteria:

* Endometriosis ≥ grade 3
* PCO syndrome
* Poor responder
* Endocrine or metabolic abnormalities

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of oocytes in both treatment groups | up to 9 months

SECONDARY OUTCOMES:
Duration of stimulation in both treatment groups, amount of gonadotropins consumed in each treatment group | up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Blockeel, MD, Principal Investigator — UZ Brussel, Centre for Reproductive Medicine, Brussels
Locations (1):
- UZ Brussel, Laarbeeklaan 101, Brussels Capital, Belgium

REFERENCES:
- [Background] Filicori M, Cognigni GE, Gamberini E, Parmegiani L, Troilo E, Roset B. Efficacy of low-dose human chorionic gonadotropin alone to complete controlled ovarian stimulation. Fertil Steril. 2005 Aug;84(2):394-401. doi: 10.1016/j.fertnstert.2005.02.036. PMID 16084880
- [Derived] Blockeel C, De Vos M, Verpoest W, Stoop D, Haentjens P, Devroey P. Can 200 IU of hCG replace recombinant FSH in the late follicular phase in a GnRH-antagonist cycle? A pilot study. Hum Reprod. 2009 Nov;24(11):2910-6. doi: 10.1093/humrep/dep253. Epub 2009 Jul 17. PMID 19617207